CLINICAL TRIAL: NCT00476047
Title: A Study of 131I-Tositumomab (Bexxar®) Consolidation in Patients With B-Cell Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma in First Remission
Brief Title: Tositumomab and Iodine I 131 Tositumomab in Treating Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma in First Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mazyar Shadman, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSOC 2301; NCI-2011-01311 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PSOC 2301 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Lymphoid Leukemia in Remission; Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage III Small Lymphocytic Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (monoclonal antibody therapy) (Experimental): Patients receive tositumomab and iodine I 131 tositumomab IV over 90 minutes on day 0 and then again 7-14 days later over 30-60 minutes.
  Interventions: Combination Product: Tositumomab and Iodine I 131 Tositumomab

INTERVENTIONS:
Combination Product: Tositumomab and Iodine I 131 Tositumomab — Give IV
  Other Names: Bexxar; Bexxar Therapeutic Regimen; Bexxar Therapy

SUMMARY:
This phase II trial studies how well tositumomab and iodine I 131 tositumomab works in treating patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) that have had their first decrease in or disappearance of signs and symptoms of cancer (first remission). Monoclonal antibodies, such as tositumomab and iodine I 131 tositumomab, may block cancer growth in different ways by targeting certain cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the progression-free survival at 2 years following administration of 131I-tositumomab (tositumomab and iodine I 131 tositumomab) in patients with CLL/SLL who achieve a complete remission (CR) or partial remission (PR) with prior therapy.

II. To improve the response rate by administering 131I-tositumomab to patients who have achieved a PR not a CR after any prior therapy.

III. To eliminate residual disease (documented by flow cytometry or polymerase chain reaction [PCR]) using 131I-tositumomab in patients who have achieved a CR after any prior therapy.

SECONDARY OBJECTIVES:

I. To evaluate the toxicities of 131I-tositumomab in 1st remission patients with previously treated CLL/SLL.

OUTLINE:

Patients receive tositumomab and iodine I 131 tositumomab intravenously (IV) over 90 minutes on day 0 and then again 7-14 days later over 30-60 minutes.

After completion of study treatment, patients are followed up weekly for 3 months, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cluster of differentiation (CD)20+ CLL/SLL; prior to the first treatment patients with CLL must have been either Rai stage III/IV disease or Rai stage I/II with evidence of disease activity as defined by the National Cancer Institute (NCI) 1996 guidelines, and patients with SLL must have been Stage III or IV per Ann Arbor staging system
* Patient has received prior therapy and is in 1st remission with a partial or complete response to treatment
* Patients must have no more than 25% of the intratrabecular marrow space involved by leukemia in bone marrow biopsy specimens as assessed microscopically after completion of treatment; bilateral posterior iliac crest core biopsies are required if the percentage of intratrabecular space involved exceeds 10% on a unilateral biopsy; the mean of bilateral biopsies must be no more than 25%
* Patient must have consented to participate in the study and signed and dated an appropriate institutional review board (IRB)-approved consent form that conforms to federal and institutional guidelines
* Patient must have a Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 (0 = fully active, able to carry on all pre-disease performance without restriction; 1 = restricted in physically strenuous activity but ambulatory and ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = ambulatory and capable of all self-care but unable to carry out any work activities and is up and about more than 50% of waking hours)
* Patient must have an anticipated survival of at least 3 months
* Granulocytes >= 1,500/uL within 14 days of planned dosimetric infusion
* Platelets >= 100,000/uL within 14 days of planned dosimetric infusion
* White blood count =< 20,000/mm^3
* Serum creatinine < 2 times upper limit of normal
* Total bilirubin < 2 times upper limit of normal
* Aspartate aminotransferase (AST) < 5 times upper limit of normal
* Males and females must agree to use a contraceptive method from enrollment to 6 months after receiving I-131 labeled tositumomab

Exclusion Criteria:

* Patients who have received prior radiolabeled antibody
* Patients with active hemolysis
* Patients must not require sustained transfusion support of blood products
* Patients in 2nd remission or beyond
* Patients who have undergone treatment with either stem cell or bone marrow transplant
* Patients with active obstructive hydronephrosis
* Patients with evidence of any significant systemic illness, active hepatitis B infection or other active infection at the time of study entry
* Patients with New York Heart Association class III or IV heart disease or other serious illness that would preclude evaluation
* Patients with known human immunodeficiency virus (HIV) infection
* Patients who are pregnant or nursing
* Patients with prior malignancy other than CLL/SLL, except for adequately treated skin cancer (basal cell or squamous cell carcinoma), in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years unless approved by the principal investigator (PI)
* Patients with active brain or leptomeningeal involvement by malignancy
* Patients who have, in the opinion of the investigator, other medical, social, or psychosocial factors that may negatively impact compliance or their safety by participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mazyar Shadman, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Monoclonal Antibody Therapy): Patients receive tositumomab and iodine I 131 tositumomab IV over 90 minutes on day 0 and then again 7-14 days later over 30-60 minutes.
  Tositumomab and Iodine I 131 Tositumomab: Give IV
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Started | 16
Completed Treatment | 16
Completed | 15
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 61 [38 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
CLL or SLL [Count of Participants; unit: Participants]
  CLL (Chronic lymphocytic leukemia) | 11
  SLL (Small lymphocytic leukemia) | 5
Prior chemotherapy [Count of Participants; unit: Participants]
  FR (fludaribine and rituximab) | 9
  FCR(fludaribine, cyclophosphamide and rituximab) | 4
  BR (bendamustine and rituximab) | 2
  R-CHOP | 1
Disease status before 131 I-tositumomab [Count of Participants; unit: Participants] — CRITERIA FOR RESPONSE Criteria for response are specified by the NCI working group guidelines; in addition, patients will be required to meet computed tomography (CT) scan criteria as defined in the protocol.
  Complete response (CR) Partial response (PR) Progressive Disease (PD) Stable Disease (SD)
  Participants
    CR (complete response) | 4
    PR (partial response) | 12
Minimal Residual Disease (MRD) status before 131 I-tositumomab [Count of Participants; unit: Participants] — MRD was assessed on bone marrow samples using 8 color flow cytometry to detect CLL/SLL cells. Any level of residual disease by flow cytometry or cytogenetics was considered MRD positive. Negativity of both tests was required to classify a patient as MRD negative.
  Participants
    Positive | 12
    Negative | 4

OUTCOME MEASURES:

1. Primary Outcome: Probability of Progression-free Survival (PFS)
Description: Progression free survival (PFS) is defined as the interval between the first treatment day to the first sign of disease progression. This outcome measures the percentage of participants with PFS at 36 months.
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 16
percentage probability | 52 [25 to 74]

2. Primary Outcome: Improved Response Rate After Treatment With 131I-tositumomab for Patients Who Had Evidence of CLL at the End of Initial Chemotherapy
Description: Response rates determined using National Cancer Institute (NCI) working group guidelines plus computed tomography (CT) scan criteria. Participants were assessed for response after initial chemotherapy and again 3 months after 131I-tositumomab treatment.Only patients who had less than a complete response (CR) after initial chemotherapy were assessed for improved response after 131I-tositumomab.
Time Frame: 3 months after 131I-tositumomab consolidation
Population: Participants who had a partial response (PR) after initial chemotherapy. Response assessed using NCI working group guidelines + CT criteria as described in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 12
Participants
  Participants who achieved a CR | 8
  Participants who did not achieve a CR | 4

3. Primary Outcome: Minimal Residual Disease (MRD) by Flow Cytometry or Polymerase Chain Reaction (PCR) in Patients Who Had a Complete Remission (CR) After Any Prior Therapy
Time Frame: 3 months after 131I-tositumomab consolidation
Measure: Count of Participants; unit: Participants
Groups:
- Patient Who Achieved CR After Any Prior Therapy: Patients who received study treatment and who had achieved a complete remission (CR) after any prior therapy.
Arm/Group | Patient Who Achieved CR After Any Prior Therapy
Number analyzed (Participants) | 4
Participants
  Negative MRD status | 4
  Positive MRD status | 0

4. Secondary Outcome: Evaluate Toxicities of 131I-tositumomab
Description: Adverse events following treatment of 131I-tositumomab
Time Frame: 48 months (median)
Measure: Number; unit: participants with this toxicity
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 16
participants with this toxicity
  Grade 3 anemia | 1
  Grade 3 or 4 neutropenia | 13
  Grade 3 or 4 thrombocytopenia | 8
  Hypogammaglobulinemia | 1
  Neutropenia related sepsis/typhlitis | 1
  Basal cell carcinoma | 2
  Squamous cell carcinoma | 1
  Myelodysplastic syndrome | 2

ADVERSE EVENTS:
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 16/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Monoclonal Antibody Therapy) (N=16)
Anemia Grade 3 (Blood and lymphatic system disorders) | 1 (1)
Neutropenia Grade 3 or 4 (Blood and lymphatic system disorders) | 13 (16)
Thrombocytopenia Grade 3 or 4 (Blood and lymphatic system disorders) | 8 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No